CLINICAL TRIAL: NCT05528952
Title: Evaluation of the Interest to Combine a CD4 Th1-inducer Cancer Vaccine Derived From Telomerase and Atezolizumab Plus Bevacizumab in Unresectable Hepatocellular Carcinoma: a Proof of Concept Randomized Phase II Study (TERTIO - Prodige 82)
Brief Title: Evaluation of the Interest to Combine a CD4 Th1-inducer Cancer Vaccine Derived From Telomerase and Atezolizumab Plus Bevacizumab in Unresectable Hepatocellular Carcinoma
Acronym: TERTIO
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: GERCOR - Multidisciplinary Oncology Cooperative Group (Other); PRODIGE (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022/680
Record Dates: First submitted 2022-09-01; First posted 2022-09-06 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Hepatocellular Carcinoma
Keywords: CD4 Th1-inducer cancer vaccine
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — atezolizumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Arm (Arm A) (Experimental): Atezolizumab + Bevacizumab + UCPVax
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab; Drug: UCPVax
- Control Arm (Arm B) (Other): Atezoliumab + Bevacizumab
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab

INTERVENTIONS:
Drug: Atezolizumab — 1200 mg IV every 3 weeks until disease progression or unacceptable toxicity
Drug: Bevacizumab — 15 mg/kg IV every 3 weeks until disease progression or unacceptable toxicity
Drug: UCPVax — UCPVax vaccine (combined with Montanide ISA51 as adjuvant) at 0.5 mg subcutaneously
  Arms: Experimental Arm (Arm A)

SUMMARY:
The TERTIO trial will propose to determine the clinical interest and immunological efficacy of a treatment combining the CD4 helper T-inducer cancer anti-telomerase vaccine (UCPVax) with anti-PD-L1 therapy (atezolizumab) and bevacizumab in unresectable HCC by evaluation of the objective response rate at 6 months (randomized phase II, 10 centers, 105 patients)

ELIGIBILITY:
Main inclusion Criteria:

1. Signed informed consent
2. Histologically confirmed hepatocellular carcinoma
3. Locally advanced, metastatic, or unresectable disease
4. Patient who had not previously received systemic anti-cancer treatment
5. Age ≥ 18 years
6. Measurable disease defined according to mRECIST guidelines (Note: Previously irradiated lesions can be considered as measurable disease only if disease progression has been unequivocally documented at that site since radiation.)
7. Patients who have received previous chemoembolization, radioembolization and/or radiotherapy should have recovered from any treatment related toxicity, to a level of ≤ grade 1 (according to National Cancer Institute [NCI] common terminology criteria for adverse events, version 5 (CTCAE v5) with the exception of Grade 2 alopecia
8. Performance status < 2
9. Child-Pugh Class A status
10. BCLC C stage or BCLC B stage not eligible to loco-regional therapy according to the Barcelona Clinic Liver Cancer (BCLC) staging system

Main exclusion Criteria:

Non-eligible to a clinical trial:

1. Patients previously exposed to anti-tumor immunotherapy as anti-PD-1, anti-PD-L1, or anti-CTLA4 agent or any immune therapy.
2. Diagnosis of additional malignancy within 3 years prior to the inclusion with the exception of curatively treated basal cell carcinoma of the skin and/or curatively resected in situ cervical or breast cancer
3. Patient with any medical or psychiatric condition or disease, which would make the patient inappropriate for entry into this study
4. Current participation in a study of an investigational agent or in the period of exclusion
5. Patient under guardianship, curatorship or under the protection of justice

   Cancer-specific exclusion criteria:
6. Know fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC
7. Uncontrolled pleural effusion, pericardial effusion, ascites or symptomatic fistula
8. Uncontrolled tumor-related pain: exposing patients to risk of exposure to corticoids or iterative hospitalizations. Symptomatic lesions amenable to palliative radiotherapy should be treated prior to inclusion. Patients should be recovered from the effects of radiation. There is no required minimum recovery period
9. Known active central nervous system metastases and/or carcinomatous meningitis. Subject with previously treated brain metastases and with radiological and clinical stability are allowed

   Non-eligible to treatment:
10. History of encephalopathy
11. Prior bleeding event due to untreated or incompletely treated esophageal and/or gastric varices within 6 months prior to randomization
12. Inadequate organ functions: known cardiac failure of unstable coronaropathy, respiratory failure, or uncontrolled infection or another life-risk condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2022-09-27 (Actual); Primary Completion 2028-03-27 (Estimated); Study Completion 2030-02-27 (Estimated)

PRIMARY OUTCOMES:
objective response rate (ORR) | at 6 months
  addition of complete response (CR) and partial response (PR) rates, evaluated by mRECIST criteria

SECONDARY OUTCOMES:
overall survival (OS) | through study completion, an average of 2 years
  delay from the date of randomization to death from any cause.
progression-free-survival (PFS) | through study completion, an average of 2 years
  delay from the date of randomization to the disease progression or death from any cause whichever occurs first
disease control rate (DCR) | at 6 months
  addition of complete response (CR), partial response (PR), and stable disease (SD) rates, evaluated by RECIST criteria v1.1 and imRECIST

CONTACTS AND LOCATIONS:
Locations (14):
- France (14):
  - CHU de Besançon, Besançon
  - CH William Morey, Chalon-sur-Saône
  - Hôpital Henri Mondor, Créteil
  - Centre Georges François Leclerc, Dijon
  - Hôpital Nord Franche-Comté, Montbéliard
  - CHU de Montpellier, Montpellier
  - CH de Mulhouse, Mulhouse
  - Institut de Cancérologie de l'Ouest, Nantes
  - Centre Hospitalier Paris St Joseph, Paris
  - Groupe Hospitalier Paris Salpetrière, Paris
  - Hôpital BEAUJON, Paris
  - Institut Mutualiste Montsouris, Paris
  - CHU de Poitiers, Poitiers
  - Hôpital Paul Brousse, Villejuif

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vienot A, Jacquin M, Rebucci-Peixoto M, Pureur D, Ghiringhelli F, Assenat E, Hammel P, Rosmorduc O, Stouvenot M, Allaire M, Bouattour M, Regnault H, Fratte S, Raymond E, Soularue E, Husson-Wetzel S, Di Martino V, Muller A, Clairet AL, Fagnoni-Legat C, Adotevi O, Meurisse A, Vernerey D, Borg C. Evaluation of the interest to combine a CD4 Th1-inducer cancer vaccine derived from telomerase and atezolizumab plus bevacizumab in unresectable hepatocellular carcinoma: a randomized non-comparative phase II study (TERTIO - PRODIGE 82). BMC Cancer. 2023 Jul 29;23(1):710. doi: 10.1186/s12885-023-11065-0. PMID 37516867